CLINICAL TRIAL: NCT05888844
Title: A Phase 2 Study Evaluating INCB099280 in Participants With Advanced Squamous Cell Carcinoma
Brief Title: A Study to Evaluate INCB099280 in Participants With Advanced Cutaneous Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 99280-212; 2022-502476-23-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: Cutaneous Squamous Cell Carcinoma; Anti-PD-L1 antibody; Metastatic cutaneous squamous cell carcinoma; Locally advanced cutaneous squamous cell carcinoma

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts. In Part 1, participants with metastatic cutaneous squamous cell carcinoma (cSCC) or locally advanced cSCC will be randomized 1:1:1 to INCB099280 Dose 1, Dose 2, or Dose 3. In Part 2, one dose level identified from Part 1 will be expanded to enroll additional participants with metastatic cSCC and locally advanced cSCC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: INCB099280 Dose 1 (Experimental): Participants will receive INCB099280 dose 1 twice daily (BID) for up to 2 years.
  Interventions: Drug: INCB099280
- Part 1: INCB099280 Dose 2 (Experimental): Participants will receive INCB099280 dose 2 twice daily (BID) for up to 2 years.
  Interventions: Drug: INCB099280
- Part 1: INCB099280 Dose 3 (Experimental): Participants will receive INCB099280 dose 3 twice daily (BID) for up to 2 years.
  Interventions: Drug: INCB099280
- Part 2: INCB099280 Dose selected from Part 1 (Experimental): Participants will receive INCB099280 dose selected from Part 1 twice daily (BID) for up to 2 years.
  Interventions: Drug: INCB099280

INTERVENTIONS:
Drug: INCB099280 — Administered as specified in the treatment arm description.

SUMMARY:
This study is being conducted to determine the safety, tolerability, and preliminary efficacy of INCB099280 in participants with advanced Cutaneous Squamous Cell Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of cSCC.
* Previously untreated or recurrent locally advanced (without nodal metastases) or metastatic (distant or regional metastasis) cSCC not amenable to curative surgery and/or radiotherapy.
* Measurable disease based on either radiographic imaging per RECIST 1.1 or WHO criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Life expectancy > 3 months.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Known history of an additional malignancy.
* Central nervous system (CNS) metastases requiring treatment and/or leptomeningeal disease.
* Toxicity from prior therapy that has not recovered.
* Prior receipt of an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent; treatment with an immune modulator (eg, CTLA-4, GITR, LAG3, TIM3, OX40, ICOS, IL-2, 4-1BB, CAR-T cell).
* Received thoracic radiation within 6 months of the first dose of study treatment.
* Participation in another interventional clinical study while receiving INCB099280.
* Impaired cardiac function or clinically significant cardiac disease.
* History or evidence of interstitial lung disease including noninfectious pneumonitis.
* Presence of gastrointestinal conditions that may affect drug absorption.
* Any autoimmune disease requiring systemic treatment in the past 5 years.
* Diagnosis of primary immunodeficiency or receiving chronic systemic steroid therapy at a daily dose exceeding 10 mg of prednisone or equivalent.
* Active infection requiring systemic therapy.
* History of organ transplantation, including allogeneic stem cell transplantation.
* Receipt of systemic antibiotics within 28 days of first dose of study treatment.
* Probiotic usage is prohibited during screening and throughout the study treatment period.
* Received a live vaccine within 28 days of the planned start of study drug.
* Laboratory values outside the Protocol-defined ranges.
* Inadequate organ function.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR), as determined by the blinded independent central review (BICR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or composite criteria for metastatic cSCC and per World Health Organization (WHO) criteria for locally advanced cSCC.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years 3 months
  Defined as any Adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug up to 90 days after the last dose of study drug or until the start of new anticancer therapy, whichever occurs first.
Number of participants with TEAEs leading to dose modification or discontinuation | Up to 2 years
  Number of participants with TEAEs leading to dose modification or discontinuation.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 2 years
  Defined as the percentage of participants with the best overall response of CR or PR, or stable disease (SD), after a minimum of 15 weeks following the initiation of study treatment as determined by the BICR per RECIST v1.1 or composite criteria for metastatic cSCC and WHO criteria for locally advanced cSCC.
Duration Of Response (DOR) | Up to 2 years
  Defined as the time from the earliest date of confirmed CR or PR to the earliest date of disease progression, as determined by the BICR according to RECIST v1.1 or composite criteria for metastatic cSCC and WHO criteria for locally advanced cSCC or death due to any cause if occurring sooner than progression.
Time to Response (TTR) | Up to 2 years
  Defined as the time from the date of first dose to the earliest date of confirmed CR or PR as determined by the BICR according to RECIST v1.1 or composite criteria for metastatic cSCC and WHO criteria for locally advanced cSCC.
Progression-free survival (PFS) | Up to 2 years
  Defined as the time from the date of first dose to the earliest date of disease progression as determined by the BICR according to RECIST v1.1 or composite criteria for metastatic cSCC and WHO criteria for locally advanced cSCC or death due to any cause if occurring sooner than progression.
Overall Survival (OS) | Up to 2 years
  Defined as the time from the date of first dose to death due to any cause.
INCB099280 pharmacokinetic (PK) in Plasma | Pre dose and 1, 2 and 6 hours post dose on Cycle 1 Day 1 and Cycle 2 Day 1. Pre dose every other cycle until Cycle 11 Day 1 (Cycle 3 Day 1, Cycle 5 Day 1, Cycle 7 Day 1, Cycle 9 Day 1 and Cycle 11 Day 1) (each cycle is 28 days)
  INCB099280 concentration in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (77):
- Australia (5):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Townsville Cancer Centre, Townsville, Queensland
  - Princess Alexandra Hospital Australia, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre Clayton, Clayton, Victoria
- Brazil (10):
  - Fundacao Pio Xii Hospital de Cancer de Barretos, Barretos
  - Cepen - Centro de Pesquisa E Ensino Em Oncologia de Santa Catarina, Florianópolis
  - Oncosite - Centro de Pesquisa Clinica E Oncologia, Ijuí
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Hospital Sao Vicente de Paulo, Passo Fundo
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hgb - Hospital Giovanni Battista - Mae de Deus Center, Porto Alegre
  - Instituto de Oncologia Saint Gallen, Santa Cruz do Sul
  - Cepho - Centro de Estudos E Pesquisas de Hematologia E Oncologia, Santo André
  - A. C. Camargo Cancer Center, São Paulo
- Canada (2):
  - Q.E. Ii Health Sciences Centre, Halifax, Nova Scotia
  - McGill University Jewish General Hospital, Montreal, Quebec
- Chile (3):
  - Cdiem - Centro de Investigacion Y Especialidades Medicas, Santiago
  - James Lind Centro de Investigacion Del Cancer, Temuco
  - Clinical Research Chile Spa., Valdivia
- Croatia (2):
  - Specialty Hospital Medico, Rijeka
  - University Hospital Centre Sestre Milosrdnice, Zagreb
- France (17):
  - Avicenne Hospital, Bobigny
  - Bordeaux Chu Hopital Saint - Andre, Bordeaux
  - Hospital Ambroise Pare, Boulogne-Billancourt
  - Chu de Clermont - Ferrand- Hospital Estaing, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Chu Dijon - Hôpital François Mitterrand, Dijon
  - Centre Hospitalier Universitaire Grenoble Alpes (Chu Grenoble Alpes) - Hopital Albert Michallon, La Tronche
  - Chru de Lille Hopital Claude Huriez, Lille
  - Chu Hopital de La Timone, Marseille
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - Chu de Nice - Hospital L Archet, Nice
  - Hospital Saint Louis, Paris
  - Centre Hospitalier de Pau - Hôpital François Mitterrand, Pau
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Charles Nicolle Chu Rouen Hospital de Bois-Guillaume, Rouen
  - University Hospital of Saint Etienne, Saint-Etienne
  - Institut Gustave Roussy, Villejuif
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Pecsi Tudomanyegyetem, Pécs
- Clinical Center of Montenegro, Podgorica, Montenegro
- Waikato Hospital, Hamilton, New Zealand
- University Clinic For Radiotherapy and Oncology, Skopje, North Macedonia
- Romania (6):
  - S.C Policlinica Ccbr S.R.L, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Medisprof, Cluj-Napoca
  - Centrul de Oncologie Sf. Nectarie Craiova, Craiova
  - S.C. Sigmedical Services Srl, Suceava
  - Oncomed Srl, Timișoara
- South Africa (6):
  - Johese Clinical Research: Midstream, Centurion
  - Chris Hani Baragwanath Hospital, Johannesburg
  - Wits Clinical Research, Johannesburg
  - The Medical Oncology Centre of Rosebank, Johannesburg
  - Phoenix Pharma (Pty) Ltd, Port Elizabeth
  - University of Pretoria Oncology Department, Pretoria
- South Korea (5):
  - Cha Bundang Medical Center, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (13):
  - Germans Trias I Pujol, Badalona
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinic Barcelona Main, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Virgen de La Arrixaca, El Palmar
  - Ico Institut Catala D Oncologia, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clinical Universidad de Navarra Madrid, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra (Cun), Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Turkey (Türkiye) (3):
  - Medical Park Seyhan Hospital, Adana
  - Ankara City Hospital, Ankara
  - Trakya University Medical Faculty, Edirne

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate INCB099280 in Participants With Advanced Cutaneous Squamous Cell Carcinoma — https://incyteclinicaltrials.com/studies/incb-99280-212